CLINICAL TRIAL: NCT02898324
Title: KiVa Anti-bullying Program in Chile: Evaluation of Effectiveness With and Without the Digital Game Component
Acronym: KiVa-Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: University of Turku (Other); Pontificia Universidad Catolica de Chile (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AKA-EDU/15
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Bullying
Keywords: Bullying; KiVa program; Primary school students
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- KiVa program full (Experimental): The schools allocated in this arm will receive the Chilean adaptation of KiVa program with all its universal and indicated actions.
  Interventions: Other: KiVa program
- KiVa program w/o the digital component (Experimental): The schools allocated in this arm will receive the Chilean adaptation of KiVa program without the digital component (online game)
  Interventions: Other: KiVa program
- Control group (No Intervention): The schools allocated in this arm will not receive the KiVa program. If successful, these schools will receive the program the following academic year.

INTERVENTIONS:
Other: KiVa program — KiVa program is an anti-bullying intervention developed in University of Turku, Finland. It is based on the participant role model, where bullying is seen as a group process focused on the bystanders' reactions to the bullying. This program includes universal and indicated actions. Universal actions include ten students lessons given by teachers where pupils learn the role of bystanders in the bullying process, how to increase empathy towards the victim, and safe strategies to supports victims. Indicated actions are delivered by a school team of three staff members, who handle acute cases of bullying.
  Arms: KiVa program full; KiVa program w/o the digital component

SUMMARY:
Bullying is a major problem worldwide and, with no exception, in Chile. Bullying is defined as a systematic aggressive behavior against a victim who cannot defend himself or herself. Victims suffer many consequences such as social isolation, psychological maladjustment, and self-injury behavior. Additionally, bullies have a higher risk for conduct problems and substance use disorders. These problems appear to last in time, affecting mental health even years later since the experience of bullying.

There are few studies in Chile aiming to determine the prevalence of bullying. In one of such studies, 47% of the students reported having been bullied during the last month before the application of the questionnaire. Even though there are many initiatives and guidelines in Chile supported by the government to help schools in order to deal with bullying, there is no any cluster randomized controlled trial (RCT) aiming to assess the effectiveness of an anti-bullying program.

KiVa anti-bullying prevention program contains universal and indicated actions. Main universal actions for 5 to 6 graders consist of 10 two-hours lessons given during a year and an online game, which have the aim to raise awareness of the role of the group in bullying, increase empathy and promote strategies to support victims. Indicated actions consist of a set of discussion groups with the victims and with the bullies with proper follow-up.

The aims of this study are: 1) To develop a culturally appropriate version of the Kiva material, and 2) to test its effectiveness of KiVa program with and without the online game, to reduce bullying behavior among low-income primary schools in Santiago using a cluster RCT design with three arms: i) KiVa full program group, ii) KiVa without online game program group, and iii) Control group.

ELIGIBILITY:
Inclusion Criteria for schools:

* Primary education
* Co-educational
* High vulnerability (measured by the Chilean index IVESINAE >75%)
* Location: Santiago, Chile.
* Exact two classes per level (5th Grade and 6th Grade), during the intervention.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4485 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Self-reported victimisation | 12 months followup
  Victimisation will be assessed using the corresponding item from the revised Olweus Bully/Victim Questionnaire (OBVQ)

SECONDARY OUTCOMES:
Self-reported bullying | 12 months followup
  Bullying actions will be assessed using the corresponding item from the revised Olweus Bully/Victim Questionnaire (OBVQ)
Peer-reported victimisation | 12 months followup
  Peer-reported victimisation will be assessed using the corresponding item from the revised Olweus Bully/Victim Questionnaire (OBVQ)
Peer-reported bullying | 12 months followup
  Peer-reported bullying will be assessed using the corresponding item from the revised Olweus Bully/Victim Questionnaire (OBVQ)
Self-reported psychological difficulties | 12 months followup
  The psychological difficulties will be assessed using the total subscale of difficulties of the Adolescent version of The Strengths and Difficulties Questionnaire (SDQ).
Self-reported psychological strengths | 12 months followup
  The psychological strengths will be assessed using the total subscale of strengths (prosocial skills) of the Adolescent version of The Strengths and Difficulties Questionnaire (SDQ).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete, MD, MSc, PhD, Principal Investigator — Universidad de Los Andes

REFERENCES:
- [Derived] Valenzuela D, Turunen T, Gana S, Rojas-Barahona CA, Araya R, Salmivalli C, Gaete J. Effectiveness of the KiVa Antibullying Program with and without the Online Game in Chile: a Three-Arm Cluster Randomized Controlled Trial. Prev Sci. 2022 Nov;23(8):1470-1482. doi: 10.1007/s11121-022-01379-z. Epub 2022 Jun 24. PMID 35739339
- [Derived] Gaete J, Valenzuela D, Godoy MI, Rojas-Barahona CA, Salmivalli C, Araya R. Validation of the Revised Olweus Bully/Victim Questionnaire (OBVQ-R) Among Adolescents in Chile. Front Psychol. 2021 Apr 12;12:578661. doi: 10.3389/fpsyg.2021.578661. eCollection 2021. PMID 33912096
- [Derived] Gaete J, Valenzuela D, Rojas-Barahona C, Valenzuela E, Araya R, Salmivalli C. The KiVa antibullying program in primary schools in Chile, with and without the digital game component: study protocol for a randomized controlled trial. Trials. 2017 Feb 20;18(1):75. doi: 10.1186/s13063-017-1810-1. PMID 28219403